CLINICAL TRIAL: NCT05615727
Title: A Randomized, Placebo-controlled Crossover Trial of Intranasal Dexmedetomidine and Zolpidem for Treatment of Primary Insomnia
Brief Title: Intranasal Dexmedetomidine and Zolpidem for Treatment of Primary Insomnia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Michael G. Irwin, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UW 21-386
Record Dates: First submitted 2022-10-12; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Insomnia
Keywords: Insomnia; Dexmedetomidine; Zolpidem
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Dexmedetomidine; Zolpidem

STUDY DESIGN:
Intervention Model Description: Each participant will take part in three sleep investigations. Each sleep investigation will take place after the participant has completed one night of sleep familiarization in the laboratory. The 3 sleep investigations will be conducted after administration of the following in a randomised manner:
  1. Placebo
  2. Intranasal dexmedetomidine
  3. Zolpidem
Who Masked: Participant, Outcomes Assessor
Masking Description: placebo-controlled crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine
- Zolpidem (Active Comparator)
  Interventions: Drug: Zolpidem
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — 2 mcg/kg of undiluted dexmedetomidine [= 0.02 ml/kg] and oral placebo tablet
  Arms: Dexmedetomidine
Drug: Zolpidem — zolpidem 10 mg and intranasal saline 0.02 ml/kg
  Arms: Zolpidem
Other: Placebo — a placebo oral tablet and intranasal saline at 0.02 ml/kg
  Arms: Placebo

SUMMARY:
Insomnia is a significant public health burden, increasing work absenteeism and health care costs in a large proportion of the population. It causes altered cognition, emotional disturbances, and reduced quality of life. The purpose of this study is to determine whether the sleep promoting effect of dexmedetomidine is superior to the conventional sleep promoting drug, zolpidem.

The main outcome of this study is to measure the time taken to fall asleep. Investigators will also look at incidences of wakening after sleep onset, sleep quality and wake time during sleep.

DETAILED DESCRIPTION:
Insomnia is a significant public health burden, increasing work absenteeism and health care costs in a large proportion of the population. It causes altered cognition, emotional disturbances, and reduced quality of life. Most epidemiologic studies have found that about one-third of adults report at least one symptom of insomnia e.g. difficulty initiating sleep or maintaining sleep. There are also similar problems related to circadian rhythm disturbance as seen in shift workers and "jet lag". Research indicates that DNA damage is apparent in doctors subjected to sleep deprivation. Traditional currently available hypnotics which are used to initiate and maintain sleep ("sleeping tablets") are either benzodiazepines (BZD) or the so-called Z-drugs (zolpidem, zopiclone and zaleplon) which are a class of psychoactive drugs that are very benzodiazepine-like in nature and act by allosterically activating gamma-aminobutyric acid receptor A (GABAA). They have virtually superseded benzodiazepines but have almost entirely the same pharmacodynamic effects and, therefore, exhibit similar action, side-effects, and risks. Despite their name, these drugs do not induce natural sleep as manifest by EEG. They are central nervous system depressants that disproportionately promote non-rapid eye movement (NREM) sleep while suppressing REM sleep. Selective REM sleep deprivation in humans has adverse effects on memory consolidation and pain perception. Other problems with these drugs include numerous reports of misuse, abuse and dependence, paradoxical reactions, increased risk of road traffic accidents and exacerbation of asthma. A retrospective cohort study of more than 100,000 age- and sex-matched patients showed that those who used these drugs were 3 times more likely to die prematurely during the 7 -year follow-up period than those who did not, with significant dose-response associations shown for benzodiazepines and the "Z drugs". New evidence-based clinical practice guidelines for the treatment of insomnia disorder were recently developed using the GRADE methodology (Grading of Recommendations, Assessment, Development, and Evaluation) and represent the first comprehensive, systematic analysis of single agents for treatment. Unfortunately, the level of evidence for all recommendations was "weak" meaning that the strength of the evidence in the published data were low. Notably, all the recommended treatments for sleep onset insomnia, besides ramelteon, a melatonin receptor agonist , are Z-drugs or BZD hypnotics. For sleep maintenance insomnia, three of five of the treatment options are Z-drugs or BZDs. The US Food and Drug Administration has recently put a Boxed Warning on Z drugs since serious injuries and death from complex sleep behaviours have occurred in patients with and without a history of such behaviours. These behaviours can occur after just one dose. Clearly, better pharmacological treatment is warranted. Dexmedetomidine is a highly selective alpha-2 adrenergic receptor antagonist that acts on the locus ceruleus1 in the brain to produce dose dependent sedation, anxiolysis and analgesia with no respiratory depression and only modest haemodynamic effects. It has been extensively studied and used for both adult and paediatric sedation, premedication, intensive care and in perioperative settings to prevent emergence delirium after anaesthesia. The sedative effect of this drug is unique in that it produces prominent slow wave activity in the electroencephalogram (EEG) resembling stage 2 NREM sleep with facilitated arousal (as with natural sleep). Of the sleeping states, the NREM sleep period seems fundamental because it happens first (wakefulness to NREM) and lasts the longest. It has even been suggested as a suitable drug to induce torpor in manned space flight. The intravenous formulation is also efficacious when administered by the intranasal route in both children and adults. Since this is not associated with any unpleasant sensation, there is increasing use for paediatric premedication and procedural sedation. The bioavailability of intranasal dexmedetomidine administered by atomiser or by drops is approximately 40% in healthy adult volunteers with an inter-individual variability of around 30%. The pharmacokinetic and pharmacodynamic profiles of the two modes of administration are similar and both are equally effective in inducing adequate sedation.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 18 to 25 years, with DSM-5 insomnia disorder. Insomnia will be diagnosed and confirmed by a clinical interview and will have an Insomnia Severity Index score of ≥ 15.

Exclusion Criteria:

1. Comorbid diagnosis of psychiatric disorders ( major depression, anxiety disorders, bipolar disorders and psychotic disorders)
2. Obstructive sleep apnoea as determined by an Apnea Hypoapnea Index of >15 or snoring.
3. Restless legs, or periodic limb movements during sleep as measured by the Periodic Limb Movements Index with arousal of > 15 per hour
4. Obesity (body mass index > 30)
5. Known or suspected cardiovascular, pulmonary, metabolic disease or diabetes as confirmed by the clinician interview during recruitment
6. Pregnancy
7. Anyone who has taken trans-meridian travel across more than one time-zone or worked night shifts in the preceding three months
8. Consuming prescribed or non-prescription sleep medication in the past month

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Sleep onset latency | 720 minutes
  Sleep onset latency is a measure of how long it takes for the participant to fall asleep once the participant gets into bed. This will be measured in minutes and reported as minutes for each of the treatments

SECONDARY OUTCOMES:
Incidence of wakening after sleep onset; Sleep quality; Wake time during sleep | 720 minutes
  Incidence of wakening after sleep onset: This is a measure of how many times the participant will wake up after falling asleep. It will be measured as count data.
  Sleep quality: This is a subjective measure and will be given as a score from a survey completed by the participant. The data will be reported as count data
  Wake time during sleep: This will be detected with the polysomnography and will be reported in total minutes

CONTACTS AND LOCATIONS:
Overall Officials: Micheal Garnet Irwin, M.B. Ch.B, Principal Investigator — The University of Hong Kong
Locations (1):
- HKU Li Ka Shing Faculty of Medicine, Hong Kong, Guangdong, China